CLINICAL TRIAL: NCT00498641
Title: Anisometropia Amblyopia Improved by Perceptual Learning and Patching
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 094-05-0112
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2007-07

CONDITIONS: Anisometropic Amblypia
Keywords: perceptual learning; occlusion therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: computer program and patching

SUMMARY:
To compare the effects of perceptual learning with patching on improving visual acuity and contrast sensitivity in payient with anisometropic amblyopia.

DETAILED DESCRIPTION:
Patients with anisometropic amblyopia were randomized to patching or perceptual learning group. Corrected amblyopic logMAR visual acuity and contrast sensitivity function were measured at four-weekly intervals until visual acuity stabilized or amblyopia resolved. Improvement in visual acuity, contrast sensitivity, and the resolution of amblyopia were compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Anisometropia without strabismus
* An interocular acuity difference of at least 0.2 logMAR in children (3-7 years of age) or in older children and adult patients without a history of patching or atropine penalization
* All patients wore their spectacle at least one year

Exclusion Criteria:

* A history of prior spectacle correction
* A history of patching or optical penalization
* The existence of an ocular disease that could contribute to decreased visual acuity
* Learning difficulties
* The presence of strabismus

Ages: 3 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Dates: Start 2005-01; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Corrected amblyopic logMAR visual acuity and contrast sensitivity function

CONTACTS AND LOCATIONS:
Overall Officials: Po Chen, MD, Study Director — Tri-Service General Hospital